CLINICAL TRIAL: NCT00878592
Title: Effect of Dietary and Life Style Modification on Post Liver Transplant Obesity
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institution
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO08010154; non applicable
Record Dates: First submitted 2009-04-08; First posted 2009-04-09 (Estimated); Last update posted 2017-10-10 (Actual); Status verified 2009-04

CONDITIONS: Post Liver Transplantation Weight Gain; Post Liver Transplantation Obesity; Nonalcoholic Steatohepatitis
Keywords: Post liver transplant; weight reduction classes; obesity; weight management; dietary and lifestyle modification
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity | interventions — Diet; Weight Reduction Programs

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (No Intervention): The first group (Group 1) will include the control subjects. They will receive one session of dietary and behavioral education.
- Dietary and Lifestyle counseling (Experimental): This group will receive a weight management and life style modification program. It consists of up to 6 weekly sessions of nutritional and physical exercise education. These initial sessions will concentrate on lifestyle modifications program including healthy food selections, emphasizing reduced fat consumption (<=30% of daily calories) and restriction of proteins to create a daily negative energy balance of ~500 kcal/day. Participants will be encouraged to start with 10 minutes of outdoor or at home physical activity such as walking or cycling then gradually increase the activity duration up to 30 minutes daily.
  Interventions: Behavioral: Dietary and life style modification

INTERVENTIONS:
Behavioral: Dietary and life style modification — This group will receive a weight management and life style modification program. It consists of up to 6 weekly sessions of nutritional and physical exercise education. These initial sessions will concentrate on lifestyle modifications program including healthy food selections, emphasizing reduced fat consumption (<=30% of daily calories) and restriction of proteins to create a daily negative energy balance of ~500 kcal/day. Participants will be encouraged to start with 10 minutes of outdoor or at home physical activity such as walking or cycling then gradually increase the activity duration up to 30 minutes daily.
  Other Names: obesity reducing regimens; besity management programs; weight reduction program
  Arms: Dietary and Lifestyle counseling

SUMMARY:
This study is to assess value of providing classes about dietary and life style modifications to decrease or prevent weight gain, less occurrence or better control of weight gain associated disorders such as high blood sugar, hypertension, heart or brain vessels problems.Candidates for this study will be those who have got liver transplant within 6 months of their post transplant period.

DETAILED DESCRIPTION:
This study is designed to be an interventional, prospective, randomized, case-control clinical trial. Procedures will be done in Starzl Transplant Institute and Center for Liver disease, Kaufmann building, UPMC.

Subjects selected to participate in this study, are adult liver transplant recipients who had undergone one liver transplantation during 6 months before the time of inclusion. They must be able to communicate in English (to be able to independently follow directives and record their activities in recall diaries). Patients will be excluded from the study if they are under 18 years old, refuse to give a written consent to participate in the study, have received liver graft more than 6 months before time of inclusion, have psychological or nervous disorders, have cardiovascular or musculoskeletal health problems interfering with basic physical activity, or have any manifestation of hepatic failure such as ascites and hepatic encephalopathy. Patients will be removed from the study if they develop intolerance to the dietary and physical recommendations (e.g. remarkable fatigue).

Verifying the eligibility of patients for participation in the study will be done through reviewing data in medical history, physical examination and investigations included in the patients' medical records. Complete blood count, liver function tests, fasting glucose and lipid profile, imaging and histopathologic investigations, abdominal imaging, pathology reports of liver biopsy, stress ECG, echocardiography. These tests are performed for standard of care.

Subjects will be randomly grouped into groups by simple randomization method. One of the investigators will randomly pick one folded paper out of a plastic bag that contains folded papers labeled on the folded side with the number of the group.

The first group (Group 1) will include the control subjects. They will receive one session of dietary and behavioral education. The second group (Group 2) will be the interventional group. They will receive a weight management and life style modification program similar to what has been previously described (Kelley et al. 2004). The program will be presented by a registered dietitian at UPMC". It consists of up to 6 weekly sessions of nutritional and physical exercise education. These initial sessions will concentrate on lifestyle modifications program including healthy food selections, emphasizing reduced fat consumption (<=30% of daily calories) and restriction of proteins to create a daily negative energy balance of ~500 kcal/day. Participants will be encouraged to start with 10 minutes of outdoor or at home physical activity such as walking or cycling then gradually increase the activity duration up to 30 minutes daily. The dietitian will provide each subject with diary for daily recording of dietary intake and physical activity respectively. Following the initial 6-week program patients will attend follow up session every 6 months for 5 years for dietary and behavioral education and to check dietary and physical activity diaries, reinforce and encourage compliance with dietary and physical exercise recommendations, answer questions and address problems. Patients will be required to attend at least 60% of the follow up sessions on site with face to face education. Attempts will be made to schedule these sessions on the same day of their regular clinical follow up to facilitate compliance. Up to 40% of monthly follow up sessions may be provided on the phone for patients who cannot attend on site because of travel restraints. The dietitian will call the candidate within few days after the missing appointment to check and encourage compliance, check for changes in weight. Each session will be held for up to 1 hour at the health education room of center for liver diseases. All sessions will be with a registered dietitian.

Additional 5 cc of blood will be taken at routine blood draws done twice in the first month then every 6 months for 5 years. The total blood volume withdrawn from each subject in both study groups is 60 cc. Blood will be spinned down, then serum will be banked in -80° Celsius freezer. These banked serum will be used in future research work aiming to assess activity of inflammatory and fibrotic markers such as tumor necrosis factor alpha, interleukin 6, leptin, and adiponectin.

Stool samples will be taken from all patients before study intervention and every 12 weeks afterwards. Stool samples will be stored at -80 degree Celsius freezer for future PCR study of fecal microflra.

Jennifer Steel will assess stress for the study candidates through specific questionnaire before start of intervention of the study and every 12 weeks afterwards.

The following data will be collected every 6 months during follow up visits for both groups; anthropometric indices of obesity such as measurements of weight, height (for BMI calculation), waist circumference, hip circumference, skin fold thickness and mid-arm circumference, survival rate, morbidity events such as cardiovascular or cerbrovascular events, diabetes and hypertension. For the control group, anthropometric measures will be obtained from them when they return for their routine clinic visits. Midarm circumference and triceps skin fold thickness will be measured to the nearest 1 cm, on the left arm midway between the tip of the acromion and the tip of olecranon. Skinfold thicknesses will be measured at triceps (Oppert et al. 2002). Waist circumference will be measured midway between iliac crest and lowest rib margin, and hip circumference at the level of the greater trochanters (Han et al. 2001).

Histological scores of necro-inflammation (Ishak score) and steatosis (Dixon's scale) of the implanted liver will be assessed at 1 year post transplant. All pathological evaluation will be done on parts (allocated for the research purpose) of biopsies obtained as deemed necessary for routine care by clinical providers (e.g. at 1 year post liver transplant) and will be conducted by the same pathologist blinded to the experimental protocol.

Data will be compared between the 2 groups by Chi square test and student t test . Assuming a rate of obesity in the control group of 50% and a 50% reduction of obesity incidence in the interventional group, we estimate that a sample size of 58 per group is needed to detect the difference with 80% confidence and a p value < 0.05. A p< 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Adult liver transplant recipients
* Those who have undergone one liver transplantation during 3 months before the time of inclusion.
* Ability to communicate in English (to be able to independently follow directives and record their activities in recall diaries).

Exclusion Criteria:

* Patients under 18 years old
* refusal to give a written consent to participate in the study
* Those who received liver graft more than 3 months before time of inclusion
* Significant cardiovascular or musculoskeletal health problems interfering with basic physical activity
* Any manifestations of hepatic failure such as ascites and hepatic encephalopathy
* Patients will be removed from the study if they develop intolerance to the dietary and physical recommendations (e.g. remarkable fatigue).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2008-10; Primary Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
waist circumference | before starting intervention, then every 6 months, afterwards for up to 5 years
weight, height (for BMI calculation) | before starting intervention, then every 6 months, afterwards for up to 5 years

SECONDARY OUTCOMES:
skin fold thickness | before starting intervention, then every 6 months, afterwards for up to 5 years
survival rate | anually for up to 5 years
Co morbidity events | anually for up to 5 years
histological scores of necro-inflammation (Ishak score) and steatosis (Dixon's scale) of the implanted liver. | at 1 year from start of inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Hossam M Kandil, MD, PhD, Principal Investigator — assistant professor of medicine
Locations (1):
- Center for Liver Diseases, UPMC., Pittsburgh, Pennsylvania, United States